CLINICAL TRIAL: NCT03535493
Title: The Effect of Acceptance and Commitment Therapy (ACT) and Float REST (Restricted Environmental Stimulation Therapy) on Burnout Syndrome.
Brief Title: The Effect of ACT and Float REST on Burnout Syndrome.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Ethics Committee concerns.
Sponsor: Amrinder Babbra (Other)
Responsible Party: Sponsor-Investigator, Amrinder Babbra, Principal Investigator, International Behavioral Research Institute
Organization: International Behavioral Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IBRI
Record Dates: First submitted 2018-05-13; First posted 2018-05-24 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Burnout Syndrome
MeSH Terms: conditions — Burnout, Psychological | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acceptance and Commitment Therapy (ACT) (Active Comparator)
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT)
- Float REST (Active Comparator)
  Interventions: Behavioral: Float REST
- ACT + Float REST (Experimental)
  Interventions: Behavioral: ACT + Float REST

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) — An ACT session entails a mindfulness-based training to foster and nurture effective behavioral and emotional responding to distress.
  Arms: Acceptance and Commitment Therapy (ACT)
Behavioral: Float REST — A float session entails laying supine in a light-proof, sound-proof tank consisting of a shallow pool of water (approximately 10 inches set to approximately 94.5 degrees to match skin temperature) with a high concentration of Epsom salt (approximately 1200 pounds) for 60 minutes.
  Other Names: Float Therapy, Isolation Tank, Sensory Deprivation Tank
  Arms: Float REST
Behavioral: ACT + Float REST — The combined intervention will combine ACT and Float REST. An ACT session entails a mindfulness-based training to foster and nurture effective behavioral and emotional responding to distress. A float session entails laying supine in a light-proof, sound-proof tank consisting of a shallow pool of water (approximately 10 inches set to approximately 94.5 degrees to match skin temperature) with a high concentration of Epsom salt (approximately 1200 pounds) for 60 minutes.
  Arms: ACT + Float REST

SUMMARY:
In 1982, Steven Hayes, a clinical psychologist, developed Acceptance and Commitment Therapy (ACT), a unique empirically based psychological intervention that uses acceptance and mindfulness strategies, together with commitment and behavior change strategies, to increase psychological flexibility. In 1954, John Lilly, a cognitive neuroscientist, developed the sensory deprivation tank (known today as Floatation Restricted Environmental Stimulation Therapy - Float REST), to access a wide range of healing, higher brain functions, and meditation through an unparalleled deep relaxation state. In this study, the investigators aim to examine whether participants in the ACT + Float REST condition will have larger decreases of the burnout phenomenon than those who receive either only ACT or Float REST.

Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
Assessing Change in Maslach Burnout Inventory - Human Services Survey (MBI-HSS) | Metric will be used as screening prior to study intervention; continuous measurement at week 2, week 4, week 6, week 8 and at one month follow-up.
  A 22 item scale that measures depersonalization, emotional exhaustion, and personal accomplishment. It is designed for professionals in human services in an array of occupations including nurses, physicians, health aides, social workers, health counselors, therapists, police, correctional officers, clergy, and other fields focused on helping people live better lives by offering guidance, preventing harm, and ameliorating cognitive, emotional, or physical problems.

CONTACTS AND LOCATIONS:
Locations (1):
- International Behavioral Research Institute, Saint Charles, Illinois, United States